CLINICAL TRIAL: NCT02173392
Title: A Bioequivalence Study Comparing a Single Subcutaneous Injection With a 1.5 mL Prefilled Syringe Versus 2 Subcutaneous Injections of 1 mL and 0.5 mL Prefilled Syringes of Brodalumab 140 mg/mL to Healthy Subjects
Brief Title: A Bioequivalence Study Comparing a Single 1.5mL Dose of Brodalumab vs. Two Doses (1.0mL + 0.5mL) of Brodalumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20130307
Record Dates: First submitted 2014-06-13; First posted 2014-06-25 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brodalumab (single 1.5mL pre-filled syringe) (Experimental): A single 210 mg subcutaneous (SC) dose of Brodalumab administered using a single 1.5mL pre-filled syringe injection
  Interventions: Drug: Brodalumab
- Brodalumab (2 pre-filled syringes [1.0mL + 0.5mL]) (Experimental): A single 210 mg subcutaneous (SC) dose of Brodalumab administered using 2 (1.0mL + 0.5mL) pre-filled syringe injections
  Interventions: Drug: Brodalumab

INTERVENTIONS:
Drug: Brodalumab — Brodalumab is a large molecule for the treatment of inflammatory diseases

SUMMARY:
A healthy subject, 2-way cross-over study to evaluate the bioequivalence of a single dose of Brodalumab vs. two doses of Brodalumab

DETAILED DESCRIPTION:
A healthy subject, 2-way cross-over study to evaluate the bioequivalence of a single 1.5mL dose of Brodalumab (140mg/mL) vs. two doses (1.0mL + 0.5mL) of Brodalumab (140mg/mL)

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females with a BMI between 18.0 and 30.0 kg/m2, inclusive. Females must be of non-reproductive potential

Exclusion Criteria:

* no history or evidence of clinically significant disorder that would pose a risk to subject safety or interfere with study evaluation, procedures, or completion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- United States (6):
  - Research Site, Glendale, California
  - Research Site, Aventura, Florida
  - Research Site, Saint Paul, Minnesota
  - Research Site, Lincoln, Nebraska
  - Research Site, Austin, Texas
  - Research Site, San Antonio, Texas

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- (Treatment A Day 1-28 + Treatment B Day 29-56): 210 mg SC Brodalumab (Single 1.5mL, Pre-filled Syringe, treatment A Days 1-28)" first, then followed by "Brodalumab (2 Pre-filled Syringes [1.0mL + 0.5mL, treatment A Days 29-56)
  Brodalumab: Brodalumab is a large molecule for the treatment of inflammatory diseases
- (Treatment B Days 1-28 + Treatment A Days 29-56): 210 mg SC Brodalumab (2 Pre-filled Syringes [1.0mL + 0.5mL, Treatment B Days 1-28])" first, then "Brodalumab (Single 1.5mL Pre-filled Syringe, treatment A Days 29-56)
  Brodalumab: Brodalumab is a large molecule for the treatment of inflammatory diseases
Period: Overall Study
Arm/Group | (Treatment A Day 1-28 + Treatment B Day 29-56) | (Treatment B Days 1-28 + Treatment A Days 29-56)
Started | 73 | 72
Completed | 59 | 68
Not Completed | 14 | 4

BASELINE CHARACTERISTICS:
Groups:
- (Treatment B Days 1-28 + Treatment 8 Days 29-56): 210 mg SC Brodalumab (2 Pre-filled Syringes [1.0mL + 0.5mL, Treatment B Days 1-28])" first, then "Brodalumab (Single 1.5mL Pre-filled Syringe, treatment A Days 29-56)
  Brodalumab: Brodalumab is a large molecule for the treatment of inflammatory diseases
- Total: Total of all reporting groups
Arm/Group | (Treatment A Day 1-28 + Treatment B Day 29-56) | (Treatment B Days 1-28 + Treatment 8 Days 29-56) | Total
Number analyzed (Participants) | 73 | 72 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (10.7) | 41.1 (10.8) | 40.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 24 | 54
  Male | 43 | 48 | 91

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameters for the Maximum Amount of Observed Brodalumab Concentration for Treatment A and Treatment B.
Description: Pharmacokinetic parameter estimates after a 210 mg dose of brodalumab, and after two 210 mg doses of brodalumab delivered subcutaneously as a single prefilled syringe (PFS) injection
Time Frame: 60 days
Population: Number of participants analyzed reflects the combination of participants analyzed at period one and then again at period two
Measure: Mean (Standard Deviation); unit: milligrams per milliliter
Groups:
- Treatment A, Brodalumab (Single 1.5mL Pre-filled Syringe): A single 210 mg subcutaneous (SC) dose of Brodalumab administered using a single 1.5mL pre-filled syringe injection
  Brodalumab: Brodalumab is a large molecule for the treatment of inflammatory diseases
- Treatment B,Brodalumab (2 Pre-filled Syringes [1.0mL + 0.5mL]): A single 210 mg subcutaneous (SC) dose of Brodalumab administered using 2 (1.0mL + 0.5mL) pre-filled syringe injections
  Brodalumab: Brodalumab is a large molecule for the treatment of inflammatory diseases
Arm/Group | Treatment A, Brodalumab (Single 1.5mL Pre-filled Syringe) | Treatment B,Brodalumab (2 Pre-filled Syringes [1.0mL + 0.5mL])
Number analyzed (Participants) | 138 | 131
milligrams per milliliter | 13.8 (7.85) | 14.8 (7.70)

2. Primary Outcome: Area Under the Drug Concentration Time Curve From Zero to the Time of Last Quantifiable Concentration of Brodalumab
Description: as for outcome 1
Time Frame: 60 days
Population: Participants analyzed is a combination of period 1 and period 2 participants results, thus the higher number of overall participants analyzed
Measure: Mean (Standard Deviation); unit: (day*mg/mL)
Arm/Group | Brodalumab (Single 1.5mL Pre-filled Syringe) | Brodalumab (2 Pre-filled Syringes [1.0mL + 0.5mL])
Number analyzed (Participants) | 138 | 131
(day*mg/mL) | 125 (69) | 149 (81.5)

3. Secondary Outcome: Immunogenicity
Description: Presence of binding or neutralizing anti-brodalumab antibodies
Time Frame: 60 days
Measure: Number; unit: participants
Arm/Group | Brodalumab (Single 1.5mL Pre-filled Syringe) | Brodalumab (2 Pre-filled Syringes [1.0mL + 0.5mL])
Number analyzed (Participants) | 141 | 131
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | (Treatment A Day 1-28 + Treatment B Day 29-56) | (Treatment B Days 1-28 + Treatment A Days 29-56)
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/131
Other Adverse Events (participants affected / at risk) | 41/141 | 39/131
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (Treatment A Day 1-28 + Treatment B Day 29-56) (N=141) | (Treatment B Days 1-28 + Treatment A Days 29-56) (N=131)
Neutropenia (Blood and lymphatic system disorders) | 4 | 3
Oropharyngeal Candidiasis (Gastrointestinal disorders) | 1 | 1
Injection Site Reaction (General disorders) | 3 | 3
Hypersensitivity (General disorders) | 1 | 6
Infections (Infections and infestations) | 10 | 10
Injection Site haemorrhage (General disorders) | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 2
Headache (Nervous system disorders) | 10 | 7
Nausea (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Muscle Strain (Musculoskeletal and connective tissue disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other